CLINICAL TRIAL: NCT04886570
Title: Clinical Follow-up of Hip Arthroplasty: A Cross-section and Longitudinal Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-05-017BC
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Hip Arthropathy; Hip Replacement
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: hip arthroplasty — Hip arthroplasty is a kind of joint reconstruction surgery, which has been successfully utilized for treatment of osteoarthritis or hip fracture for decades. In this surgery, implants is applied to reconstruct hip joint, and usually comprised of four components, including femoral stem, femoral head, acetabular cup and liner.

SUMMARY:
This longitudinal follow-up study aims to analyze how surgical and patient characteristics affect clinical outcomes in the subjects received total hip arthroplasty (THA) or hemiarthroplasty (HA).

DETAILED DESCRIPTION:
Clinical assessments in this research include visual analogue scale (VAS), Harris Hip Score (HHS), Oxford Hip Score (OHS), forgotten joint score (FJS-12) and X-ray imaging applied to examine the stability of implants. Through analyzing surgical information, functional measures and self-reported questionnaires, this study intends to gain insights into the correlations between various clinical aspects.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years old at least.
2. Osteoarthritis (OA)
3. Avascular necrosis
4. Rheumatoid arthritis (RA)
5. Previous failure of hemiarthroplasty
6. Femoral head or neck or trochanteric fractures
7. Developmental dysplasia of the hip

Exclusion Criteria:

1. Being unable or unwilling to participate in
2. Subjects having cognitive impairment cannot fill out survey
3. Other complication causing severe deficiency in function and motion

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects receiving hip arthroplasty in Taipei Veterans General Hospital meet the inclusion criteria can be considered to recruit
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Pre-operation, 6 weeks, 12 weeks and 1 year after surgery
  Visual Analogue Scale (VAS) is a patient-reported outcome measure. Scale from 0 to 10 stands for no pain to extreme pain.
Harris Hip Score | Pre-operation, 6 weeks, 12 weeks and 1 year after surgery
  Harris Hip Score (HHS) assesses the results of hip replacement. the domains cover pain, function, absence of deformity and range of motion. The maximum score of HHS is 100, and the higher score participants get, the less dysfunction they have.
Oxford Hip Score | Pre-operation, 6 weeks, 12 weeks and 1 year after surgery
  Oxford Hip Score (OHS) is a patient-reported outcome measure with 12 questions related to the condition of function and pain. Total scores is from 0 to 48, higher scores represent a better outcome.
Forgotten Joint Score (FJS-12) | Pre-operation, 6 weeks, 12 weeks and 1 year after surgery
  Forgotten Joint Score (FJS-12) is a patient-reported questionnaire with 12 questions, assessing the ability of the patient to forget the affected joints during daily activities. The higher the scores, the better the outcome.
Radiographic analysis | Pre-operation, 6 weeks, 12 weeks and 1 year after surgery
  X-ray imaging will be applied to examine the stability of implants, such as radiolucent line and loosening. The width of radiolucent line around implant suggest the possibility of implant loosening; generally, the wider the width is, the higher risk of loosening.

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Szu Yang, Principal Investigator — Department of orthopedics, Taipei Veterans General Hospital, Taipei, Taiwan